CLINICAL TRIAL: NCT03623620
Title: Preventing Depressive Relapse in Pregnant Women With Recurrent Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Colorado, Boulder (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Lee S. Cohen, MD, Director, Center for Women's Mental Health, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018P001472; R01MH117253 (NIH)
Record Dates: First submitted 2018-08-02; First posted 2018-08-09 (Actual); Results first posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: Depression; Pregnancy Related; Antenatal Depression
Keywords: Depression; Pregnancy; Antidepressants; Mindfulness; Medication use during pregnancy; Depression Relapse; Suicidal ideation
MeSH Terms: conditions — Depression; Suicidal Ideation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital delivery of MBCT (Mindful Mood Balance for Moms) (Experimental): Subjects will receive digital delivery of mindfulness-based cognitive therapy (Mindful Mood Balance for Moms) for 12 weeks, along with the usual care they would receive from their provider.
  Interventions: Behavioral: Digital Delivery of Mindfulness-Based Cognitive Therapy
- Usual Care (No Intervention): Subjects will receive only usual care, the care they would normally receive from their community provider, for 12 weeks.

INTERVENTIONS:
Behavioral: Digital Delivery of Mindfulness-Based Cognitive Therapy — 12-week program that emphasizes mindfulness and cognitive behavioral skills
  Arms: Digital delivery of MBCT (Mindful Mood Balance for Moms)

SUMMARY:
The purpose of this investigation is to conduct a pragmatic effectiveness trial comparing digital mindfulness-based cognitive therapy (MBCT) plus usual care to usual care (UC) only among euthymic pregnant women with recurrent depression treated with antidepressants.

In the supplemental arms we will investigate the prevalence, severity, longitudinal course, correlates, and predictors of suicidal ideation and behavior among women during pregnancy and the postpartum period.

DETAILED DESCRIPTION:
This study will address a significant gap in the evidence regarding effective approaches to prevent depressive relapse among women with recurrent depression who maintain euthymia using antidepressants and who wish to conceive or who are pregnant. Relapse rates of depression following antidepressant discontinuation among such women has been established, and the efficacy of MBCT in mitigating relapse risk in pregnant women with recurrent depression compared to UC also has been demonstrated. But the effectiveness of MBCT has not been tested in a definitive trial; the question of whether MBCT can mitigate risk for depressive relapse among pregnant women on antidepressants, including among those who discontinue antidepressants proximate to or during pregnancy, also has not been addressed.

Reproductive age women with recurrent depression and their healthcare providers need to know, first, if a scalable digital non-pharmacologic prevention approach is superior to UC in community settings, and second, whether MBCT can attenuate risk for depressive relapse among those who elect to discontinue maintenance antidepressant treatment proximate to or during pregnancy. Lastly, the capacity to identify which women are most likely to benefit from a non-pharmacologic or pharmacologic approach personalizes the risk benefit decision making process for reproductive age women on antidepressants planning to conceive or who are pregnant.

Investigators will test the relative risk for depressive relapse and reduction of symptom burden between women randomized to digital MBCT or UC, explore the specific benefit of MBCT relative to antidepressant discontinuation, and determine whether a treatment selection algorithm can predict whether MBCT or UC will work best for a specific participant.

The supplemental arms of this study will further investigate suicidal ideation and behavior in a perinatal population to better understand the prevalence, severity, longitudinal course, correlates and predictors of suicidal ideation and behavior among women during pregnancy and in the postpartum period.

Investigators will use a mixed methods approach of both cross-sectional and longitudinal study designs to characterize a real-world population of pregnant and postpartum women who have endorsed suicidality. Investigators will also use qualitative interviews, self-report instruments, and medical records to explore the extent to which community healthcare professionals providing care to perinatal women report the knowledge base and requisite skills to address suicidal ideation and behavior in this population.

MMB for Moms delivers digitally both the content and structure of in-person MBCT, and may be a promising intervention for pregnant women with suicidal ideation. Investigators will also explore the safety, feasibility, and acceptability of enrolling pregnant women with any reports of suicidal ideation or behavior in a proof of concept randomized controlled trial comparing MMB for Moms to enhanced usual care.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Ages 18 or older
* History of recurrent major depression prior to pregnancy (at least 2 prior episodes, one of which may be currently treated)
* Euthymic or with residual symptoms (PHQ-9 ≤ 9)
* No depressive relapse since last menstrual period
* Currently or recently received antidepressants (within the three months prior to last menstrual period)
* Presence of ongoing community provider

Exclusion Criteria:

* Diagnosis of bipolar or psychotic disorder
* Active mania, psychosis, or substance abuse (within the last 6 months)
* Immediate risk of self-harm
* Non-English speaking

Inclusion and exclusion criteria for the participants in the supplemental arms of the study differ from the main study and are as follows:

Arm 1 Aim 1a

Inclusion Criteria:

* Pregnant women (prior to 16 weeks gestation)
* Age 18 or older
* Presence of an ongoing community prescriber / provider
* Suicidal ideation as noted by item #9 of the PHQ-9
* History of recurrent depression, dysthymia or subsyndromal depression

Exclusion Criteria:

* Diagnosis of bipolar or psychotic disorder
* Mania, psychosis, or active substance abuse (within the last 6 months for substance abuse)
* Non-English speaking

Arm 1 Aim 1b

Inclusion Criteria:

* Age 18 or older
* Current prenatal healthcare provider of a participant enrolled in Arm 1 Aim 1a

Exclusion Criteria:

* Non-English speaking

Arm 1 Aim 1c

Inclusion Criteria:

* Pregnant women
* Age 18 or older
* Self-reported history of major depressive disorder
* Suicidal ideation as noted by item #9 of the PHQ-9

Exclusion Criteria:

* Non-English speaking

Arm 2

Inclusion Criteria:

* Pregnant women (prior to 16 weeks gestation)
* Age 18 or older
* History of recurrent major depression prior to pregnancy (at least two prior episodes, one of which may be currently treated)
* Euthymic or with residual symptoms (PHQ-9 </=9)
* Presence of an ongoing community prescriber / provider
* Current suicidal ideation as noted by item #9 of the PHQ-9 or past suicidal ideation as noted by item A3g on the MINI mood module

Exclusion Criteria:

* Diagnosis of bipolar or psychotic disorder
* Mania, psychosis, or active substance abuse (within the last 6 months for substance abuse)
* Non-English speaking

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females
Enrollment: 500 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee S Cohen, MD, Principal Investigator — Massachusetts General Hospital; Sona Dimidjian, PhD, Principal Investigator — University of Colorado, Boulder
Locations (2):
- United States (2):
  - University of Colorado Boulder, Boulder, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared via the National Database for Clinical Trials related to Mental Illness (NDCT) every 6 months after enrollment begins, and before publication. In addition, de-identified data and accompanying documentation describing and referencing all variables will be available for use by other investigators upon request.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will become available 6 months after study start-up and will continue to be available throughout the study.
Access Criteria: Interested investigators will be asked to submit a proposal form, which will be reviewed by the principal investigator for scientific integrity and adherence to ethical guidelines.

REFERENCES:
- [Background] Cohen LS, Altshuler LL, Harlow BL, Nonacs R, Newport DJ, Viguera AC, Suri R, Burt VK, Hendrick V, Reminick AM, Loughead A, Vitonis AF, Stowe ZN. Relapse of major depression during pregnancy in women who maintain or discontinue antidepressant treatment. JAMA. 2006 Feb 1;295(5):499-507. doi: 10.1001/jama.295.5.499. PMID 16449615
- [Background] Dimidjian S, Goodman SH, Felder JN, Gallop R, Brown AP, Beck A. Staying well during pregnancy and the postpartum: A pilot randomized trial of mindfulness-based cognitive therapy for the prevention of depressive relapse/recurrence. J Consult Clin Psychol. 2016 Feb;84(2):134-45. doi: 10.1037/ccp0000068. Epub 2015 Dec 14. PMID 26654212

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The UPWARD randomized clinical trial was conducted nationally, recruiting euthymic pregnant women with recurrent depression treated with antidepressants. Participant recruitment for UPWARD began March 7, 2019, and concluded July 8, 2020.
Pre-assignment Details: 745 individuals were eligible after the initial phone screen, 512 completed the baseline interview and surveys (66 were found ineligible during the baseline interview, 20 did not complete baseline surveys within 1 week, and 147 were non-responsive to follow-up), and 500 were randomized (12 were lost to follow up before randomization).
Period: Overall Study
Arm/Group | Digital Delivery of MBCT (Mindful Mood Balance for Moms) | Usual Care
Started | 249 | 251
Completed | 249 | 251
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Digital Delivery of MBCT (Mindful Mood Balance for Moms) | Usual Care | Total
Number analyzed (Participants) | 249 | 251 | 500
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 249 | 251 | 500
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.1 (4.65) | 32.2 (4.43) | 32.2 (4.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 249 | 251 | 500
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 29 | 46
  Not Hispanic or Latino | 232 | 222 | 454
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 8 | 9 | 17
  Native Hawaiian or Other Pacific Islander | 3 | 2 | 5
  Black or African American | 11 | 14 | 25
  White | 216 | 210 | 426
  More than one race | 5 | 9 | 14
  Unknown or Not Reported | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Relapse of Depression
Description: Depression relapse from randomization through 6 month postpartum
Time Frame: Randomization through 6 months postpartum
Measure: Number; unit: Participants
Arm/Group | Digital Delivery of MBCT (Mindful Mood Balance for Moms) | Usual Care
Number analyzed (Participants) | 249 | 251
Participants | 81 | 111

ADVERSE EVENTS:
Time Frame: March 12, 2019 to September 12, 2021 (18 months)
Description: Adverse events were probed for in every phone interview with study participants using standardized health questionnaires for each interview timepoint.
Arm/Group | Digital Delivery of MBCT (Mindful Mood Balance for Moms) | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/249 | 0/251
Serious Adverse Events (participants affected / at risk) | 0/249 | 0/251
Other Adverse Events (participants affected / at risk) | 177/249 | 209/251
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Digital Delivery of MBCT (Mindful Mood Balance for Moms) (N=249) | Usual Care (N=251)
All events categorized as "unexpected" and "non-Severe" (Pregnancy, puerperium and perinatal conditions) | 177 (177) | 209 (209) — Any non-severe, unexpected, and non-study related complications occurring during the perinatal period (ex: placenta problems, gestational diabetes, eclampsia/pre-eclampsia, pre-term labor/delivery, breech/abnormal fetal presentation, etc.)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-17): https://cdn.clinicaltrials.gov/large-docs/20/NCT03623620/Prot_SAP_000.pdf